CLINICAL TRIAL: NCT01784159
Title: Impact of Aspirin Use on the Severity of Organ Dysfunctions in Patients With Sepsis and Septic Shock: a Randomized, Double-blind, Placebo-controlled Trial - ASP-SEPSIS.
Brief Title: ASpirin for Patients With SEPsis and SeptIc Shock
Acronym: ASP-SEPSIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated: The study was stopped prematurely and will not be resumed due to the higher number of bleeding cases in the intervention group, as recomended by the Data Safety Monitoring Board on February 7, 2023.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Flavia Ribeiro Machado, Professor of Intensive Care Medicine, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPM81449
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Sepsis
Keywords: ICU; Sepsis; Aspirin; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 1tb / day/ 7days
  Interventions: Drug: Aspirin
- Aspirin (Active Comparator): Intervention aspirin 200 mg/day for 7 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin administration for 7 days
  Other Names: AAS

SUMMARY:
This Randomized, pragmatic, multicentric with blinding of patients and health professionals, intention-to-treat analysis has by primary endpoint to evaluate whether the aspirin use reduces the intensity of organic dysfunction measured by the variation of the SOFA score starting from the day of admission to the seventh day. Secundary endpoint: To evaluate if the aspirin use reduces the time of mechanical ventilation, length of stay in the ICU and in the hospital. In addition, to evaluate the safety of its administration regarding the occurrence of bleeding.

The data will be collected directly from the chart of the patients admitted to the ICU.

Data quality assurance will be made through periodic verification, aiming for complete and consistent data. The centers will receive periodic reports for adequacy of potentially inconsistent or incomplete data.

The baseline SOFA of patients with sepsis is 8.8 with a standard deviation of 3. The expected reduction in the control group in the SOFA at day 7 is 2 points. Considering a power of 80% and a level of significance of 0.05, it is estimated that 109 patients will be needed in each group. A total of 218 patients will compose the sample.

All analyzes will follow the intention-to-treat principle. We will evaluate the effect of aspirin compared to placebo on primary and binary outcomes by means of relative risks, 95% confidence intervals and chi-square tests. For continuous outcomes with normal distribution, we will present the mean difference, 95% confidence interval and P value calculated by t test. For continuous outcomes with asymmetric distribution, we will perform Wilcoxon test.

DETAILED DESCRIPTION:
Design Randomized, pragmatic, multicentric with blinding of patients and health professionals.

Bias control Allocation secrecy with web randomization. Blinding of patients and health professionals. Intention-to-treat analysis.

Primary endpoint To evaluate whether the aspirin use reduces the intensity of organic dysfunction measured by the variation of the SOFA score starting from the day of admission to the seventh day.

Secondary endpoint To evaluate if the aspirin use reduces the time of mechanical ventilation, time with vasopressors, time in renal replacement therapy, length of stay in the ICU and in the hospital. In addition, to evaluate the safety of its administration regarding the occurrence of bleeding.

Eligibility

Inclusion criteria:

The three criteria below must be present:

1. Signature of informed consent
2. Patients must be older than 18 years old
3. Diagnosis of sepsis and/or septic shock for less than 48 hours with at least one of the following organ dysfunctions:

   * Lactate above 4mmol/L (36mg/dL)
   * Thrombocytopenia < 100,000/mm3 or reduction > 50% in the count in the last 3 days
   * PaO2/FiO2 < 200 without signs of apparent volume overload
   * Hypotension MAP < 65mmHg refractory to volume replacement with the need to use vasopressor

Exclusion Criteria:

1. Pregnancy
2. Impossibility to use the intestinal tract
3. Death perspective in less than 24 hours
4. Patients in the end of their lives or in exclusive palliative care
5. Patients with active bleeding
6. Prior study participation
7. Known allergy to aspirin
8. Active peptic ulcer
9. Previous use of antiplatelet agents in the last 7 days
10. Previous use of AINEs in the last 7 days, except for dipyrone.
11. Hemorrhagic stroke in the last 7 days or central nervous system surgery in the last 72 hours.
12. Platelets <30,000 cells/mm3.
13. Large surgery in the last 24 hours if the attending surgeon judges that the risk of bleeding is high enough that aspirin cannot be used.
14. Ophthalmologic surgery postoperative and transurethral resection of the prostate at the discretion of the attending physician.
15. Hepatic cirrhosis or previous liver disease with altered prothrombin activity, manifested by INR above 2.0 or other previous coagulopathies.
16. Severe head injury in the last 7 days.
17. Use or indication of anticoagulation.

Study intervention The treatments to be compared in the study are a dose of 200 mg of aspirin daily for 7 days and placebo. Both look identical.

Study outcomes

Primary outcomes:

• Variation of the SOFA score between D7 and D1

Secondary outcomes:

* Death in the ICU
* Days free of mechanical ventilation within 28 days
* Days free of vasopressor within 28 days
* Length of ICU stay
* Length of hospital stay
* Renal injury KDIGO >= 2 within 7 days
* Renal replacement therapy use
* Major bleeding occurency
* Count of unitis of red blood cells received in 14 days

Data management The data will be collected directly from the chart of the patients admitted to the ICU. Data quality assurance will be made through periodic verification, aiming for complete and consistent data. The centers will receive periodic reports for adequacy of potentially inconsistent or incomplete data.

Statistics The baseline SOFA of patients with sepsis is 8.8 with a standard deviation of 3. The expected reduction in the control group in the SOFA at day 7 is 2 points. Considering a power of 80% and a level of significance of 0.05, it is estimated that 109 patients will be needed in each group. A total of 218 patients will compose the sample.

ELIGIBILITY:
Eligibility - patients:

Inclusion criteria:

The three criteria below must be present:

1. Signature of informed consent
2. Patients must be older than 18 years old
3. Diagnosis of sepsis and/or septic shock for less than 48 hours with at least one of the following organ dysfunctions:

   * Lactate above 4mmol/L (36mg/dL)
   * Thrombocytopenia < 100,000/mm3 or reduction > 50% in the count in the last 3 days
   * PaO2/FiO2 < 200 without signs of apparent volume overload
   * Hypotension MAP < 65mmHg refractory to volume replacement with the need to use vasopressor
   * Acute renal injury increased by 2.0 to 2.9 times from baseline or diuresis rate less than 0.5ml/kg/h for more than 12 hours

Exclusion Criteria:

1. Pregnancy
2. Impossibility to use the intestinal tract
3. Death perspective in less than 24 hours
4. Patients in the end of their lives or in exclusive palliative care
5. Patients with active bleeding
6. Prior study participation
7. Known allergy to aspirin
8. Active peptic ulcer
9. Previous use of antiplatelet agents in the last 7 days
10. Previous use of AINEs in the last 7 days, except for dipyrone.
11. Hemorrhagic stroke in the last 7 days or central nervous system surgery in the last 72 hours.
12. Platelets <30,000 cells/mm3.
13. Large surgery in the last 24 hours if the attending surgeon judges that the risk of bleeding is high enough that aspirin cannot be used.
14. Ophthalmologic surgery postoperative and transurethral resection of the prostate at the discretion of the attending physician.
15. Hepatic cirrhosis or previous liver disease with altered prothrombin activity, manifested by INR above 2.0 or other previous coagulopathies.
16. Severe head injury in the last 7 days.
17. Use or indication of anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Difference between the Sequential Organ Failure Assessment (SOFA) Score on the seventh day of ICU stay and baseline (DeltaSOFA D7-D1). | 7 days
  To evaluate whether the aspirin use reduces the intensity of organic dysfunction. measured by the variation of the SOFA score starting from the day of admission to the seventh day. The Sequential Organ Failure Assessment (SOFA) Score ranges between 0 and 24.

SECONDARY OUTCOMES:
Mechanical ventilation free days; | 28 days
  To evaluate if the aspirin use reduces the time of mechanical ventilation, that ranges between 0 and 28 days.
Vasopressor free days | 28 days
  To evaluate if the aspirin use reduces the days using vasoressors, that ranges between 0 and 28 days.
Intensive Care Unit (ICU) free days | 28 days
  Length of stay in the ICU, that ranges between 0 and 28 days
Hospital free days | 28 days
  Length of stay in the hospital, that ranges between 0 and 28 days
Renal replacement therapy | 28 days
  Length of stay in renal replacement therapy, that ranges between 0 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Machado, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Almeida TML, Freitas FGR, Figueiredo RC, Houly SG, Azevedo LCP, Cavalcanti AB, Damiani LP, Svicero BS, Souza MA, Bustamante CLS, Ramos FJS, Alves RSV, Atallah FC, Jackiu M, Pacheco ES, Schmidt RC, Serra FSC, Tomotani DYV, Zampieri FG, Machado FR; BRICNET. Acetylsalicylic Acid Treatment in Patients With Sepsis and Septic Shock: A Phase 2, Placebo-Controlled, Randomized Clinical Trial. Crit Care Med. 2025 Feb 1;53(2):e269-e281. doi: 10.1097/CCM.0000000000006564. Epub 2025 Feb 21. PMID 39982179